CLINICAL TRIAL: NCT05859581
Title: To Explore the Value of Colon MRI in Assessing the Status of Retroperitoneal Resection Margin Following Beyond Complete Mesocolic Excision Surgery for Advanced Colon Cancer
Brief Title: The Value of MRI in Assessing the Status of Retroperitoneal Resection Margin in Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Colon MRI-2023-01
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Colon Cancer
Keywords: Colon cancer; MRI; Resection margin
MeSH Terms: conditions — Colonic Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected positive RPRM on MRI (Experimental)
  Interventions: Procedure: Beyond complete mesocolic excision surgery

INTERVENTIONS:
Procedure: Beyond complete mesocolic excision surgery — If the participants were diagnosed with positive retroperitoneal resection margin (RPRM), they underwent beyond complete mesocolic excision surgery to ensure the R0 resection.

SUMMARY:
The goal of this clinical trial is to explore the value of colon MRI in assessing the status of retroperitoneal resection margin (RPRM) for advanced colon cancer.

The main questions it aims to answer are:

* Concordance between MRI suspected RPRM positive and pathologically confirmed positive.
* Can RPRM-positive patients undergo beyond complete mesocolic excision (CME) surgery in order to achieve R0 resection?

Participants will undergo colon MRI examination and once MRI suspects RPRM positive, they will receive beyond CME surgery.

ELIGIBILITY:
Inclusion Criteria:

* primary colon adenocarcinoma confirmed by biopsy
* preoperative CT suspecting retroperitoneal resection margin (RPRM) positive
* received colon MRI scan
* underwent beyond complete mesocolic excision surgery
* sufficient clinical and pathological results

Exclusion Criteria:

* combined with other malignant tumors
* simultaneous distant metastasis
* definite invaded other organs or structures (T4b tumors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Coincidence rate with pathological result | within 2 weeks after surgery
  Coincidence rate between MRI diagnosed retroperitoneal resection margin and pathologically confirmed positive

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Shi Sun, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No